CLINICAL TRIAL: NCT06297577
Title: Clinical Evaluation of Injectable Albumin Platelet Rich Fibrin (Alb-PRF) Versus Minimally Invasive Surgical Technique (MIST) in the Management of Intra-bony Defect in Stage-III Periodontitis Patients. A Randomized Controlled Clinical Trial
Brief Title: Clinical Evaluation of Injectable Alb-PRF in the Management of Intrabony Defect in Stage-III Periodontitis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mashaal Mohammed Abdullah Mohammed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MASH2024
Record Dates: First submitted 2024-02-18; First posted 2024-03-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Intrabony Periodontal Defect
Keywords: Albumin Platelet Rich Fibrin (Alb-PRF); Minimally Invasive Surgical Technique (MIST); Stage 3 periodontitis; Intrabony defect
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the type of intervention, only the outcome assessor and the statistician will be blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Albumin Platelet Rich Fibrin (Alb-PRF) (Experimental): For the production of Alb-PRF membrane, two 10 ml vacuum plastic tubes will be centrifuged at 700 g for 8 minutes. After centrifugation, the upper layer (yellow layer) shows the liquid plasma layer. The most upper layer of platelet-poor plasma (PPP) will be collected in a syringe and then will be heated in a heat block device at 75°C for 10 minutes to create denatured albumin (albumin gel). After heating, the albumin gel will be cooled to room temperature for approximately 10 minutes. An injectable albumin gel was then prepared. The liquid platelet-rich layer (liquid-PRF), including the buffy coat layer with accumulated platelets, leukocytes and growth factors, will be collected in a separate syringe and will be reserved at room temperature (20°C). The albumin gel and liquid PRF will be then thoroughly mixed by utilizing a female-female luer lock connector
  Interventions: Procedure: Albumin Platelet Rich Fibrin (Alb-PRF) combined with minimally invasive surgical technique (MIST)
- Minimally Invasive Surgical Technique (MIST) (Active Comparator): Surgical approach will be the Minimally Invasive Surgical Technique (MIST) approach according to; simplified or modified papilla-preservation flap design upon the papilla width.
  Defects will be thoroughly debrided using Gracey curettes and ultrasonic scalers.
  Then, a single internal mattress suture using 5-0 polypropylene sutures will be placed at the defect-associated inter-dental area.
  Interventions: Procedure: Minimally invasive surgical technique (MIST)

INTERVENTIONS:
Procedure: Albumin Platelet Rich Fibrin (Alb-PRF) combined with minimally invasive surgical technique (MIST) — Albumin-PRF will be placed into intrabony defect
  Arms: Albumin Platelet Rich Fibrin (Alb-PRF)
Procedure: Minimally invasive surgical technique (MIST) — MIST will be the surgical access for treatment of Intrabony defect
  Arms: Minimally Invasive Surgical Technique (MIST)

SUMMARY:
Clinical Evaluation of Injectable Albumin Platelet Rich Fibrin Versus Platelet Rich Fibrin in the Management of Intra-bony Defect in Stage-III Periodontitis Patients.

The goal of this clinical trial is to compare Injectable Albumin Platelet Rich Fibrin Versus Platelet Rich Fibrin in the Management of Intra-bony Defect in Stage-III Periodontitis Patients. The main question aims to answer are:

will Albumin Platelet Rich Fibrin (Alb-PRF) as adjunct to minimally invasive surgical technique (MIST) be superior in terms of improvement in clinical parameters compared to the use of PRF with MIST.

ELIGIBILITY:
Inclusion Criteria:

1. Stage III periodontitis patient having at least one tooth with 2-wall, 3-wall, or combined 2- to 3-wall intrabony defect ≥3 mm in depth (assessed by bone sounding, radiographic examination) with clinical attachment level (CAL) ≥5mm and probing pocket depth (PPD) ≥6 mm with no defect extending to a root furcation area.
2. Vital teeth.
3. No history of intake of antibiotics or other medications affecting the periodontium in the previous 6 months.
4. No periodontal therapy carried out in the past 6 months.
5. Ability to sign an informed consent form.
6. Patients age ≥18 years old.
7. Patients who are cooperative, motivated, and hygiene conscious.
8. Systemically free according to Cornell Medical Index.

Exclusion Criteria:

1. Patient undergoing orthodontic treatment.
2. Pregnant females or breast feeding.
3. Smokers.
4. Teeth mobility greater than grade I.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-08-30 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level (CAL) | CAL will be measured at base line, 6, and 9 months postoperative
  CAL will be measured from the cemento-enamel junction to the bottom of the gingival sulcus/periodontal pocket using the University of North Carolina periodontal probe at six sites per tooth.

SECONDARY OUTCOMES:
Probing Depth (PD) | CAL will be measured at base line, 6, and 9 months postoperative
  PD will be measured from the gingival margin to the bottom of the gingival sulcus/ periodontal pocket using the University of North Carolina periodontal probe at six sites per tooth.
Radiographic Linear Defect Depth (RLDD) | Radiographic defect fill will be measured at base line, 6, and 9 months postoperative
  Individually customized bite blocks will be fabricated for each patient and parallel-angle technique will be employed using X-ray film holding system. Periapical radiograph PSP sensor size two and standardized exposure setting of 60 kVp, 8 mA, 0.7 mm, and 0.10 s will be used. RLDD will be measured as the depth of the intrabony defect from the alveolar crest (AC) to the defect base (DB)
Recession Depth (RD) | RD will be measured at base line, 6, and 9 months postoperative
  RD will be measured from the cemento-enamel junction to the most apical extension of the gingival margin using the University of North Carolina periodontal probe at six sites per tooth.
Post-operative Pain | During first week postoperative
  The visual analogue scale (VAS) score (0-10)
Radiographic defect fill (RDF) | Radiographic defect fill will be measured at base line, 6, and 9 months postoperative
  Calculation of bone fill in mm will be done by a subtraction of follow-up from baseline RLDD values

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hosny, Professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No
starting 6 months after publication

REFERENCES:
- [Result] Fujioka-Kobayashi M, Schaller B, Mourao CFAB, Zhang Y, Sculean A, Miron RJ. Biological characterization of an injectable platelet-rich fibrin mixture consisting of autologous albumin gel and liquid platelet-rich fibrin (Alb-PRF). Platelets. 2021 Jan 2;32(1):74-81. doi: 10.1080/09537104.2020.1717455. Epub 2020 Jan 20. PMID 31959025
- [Result] Miron RJ, Chai J, Fujioka-Kobayashi M, Sculean A, Zhang Y. Evaluation of 24 protocols for the production of platelet-rich fibrin. BMC Oral Health. 2020 Nov 7;20(1):310. doi: 10.1186/s12903-020-01299-w. PMID 33160335
- [Result] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S173-S182. doi: 10.1002/JPER.17-0721. PMID 29926951
- [Result] Pavlovic V, Ciric M, Jovanovic V, Trandafilovic M, Stojanovic P. Platelet-rich fibrin: Basics of biological actions and protocol modifications. Open Med (Wars). 2021 Mar 22;16(1):446-454. doi: 10.1515/med-2021-0259. eCollection 2021. PMID 33778163
- [Result] Alshoiby MM, Fawzy El-Sayed KM, Elbattawy W, Hosny MM. Injectable platelet-rich fibrin with demineralized freeze-dried bone allograft compared to demineralized freeze-dried bone allograft in intrabony defects of patients with stage-III periodontitis: a randomized controlled clinical trial. Clin Oral Investig. 2023 Jul;27(7):3457-3467. doi: 10.1007/s00784-023-04954-y. Epub 2023 Mar 31. PMID 37002441
- [Result] Gheno E, Mourao CFAB, Mello-Machado RC, Stellet Lourenco E, Miron RJ, Catarino KFF, Alves AT, Alves GG, Calasans-Maia MD. In vivo evaluation of the biocompatibility and biodegradation of a new denatured plasma membrane combined with liquid PRF (Alb-PRF). Platelets. 2021 May 19;32(4):542-554. doi: 10.1080/09537104.2020.1775188. Epub 2020 Jun 12. PMID 32531175